CLINICAL TRIAL: NCT03111316
Title: Combined Use of the Controlled Release Dinoprostone Insert and Foley Catheter Compared to the Foley Catheter Alone for Cervical Ripening and Labor Induction in Term Women: A Randomized Controlled Trial
Brief Title: Foley Catheter Compared to the Foley Catheter Alone for Cervical Ripening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ferring
Record Dates: First submitted 2017-03-13; First posted 2017-04-12 (Actual); Results first posted 2019-05-03 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Cervical Ripening; Induction of Labor
Keywords: Cervical Ripening; Induction of Labor
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Foley Catheter & Dinoprostone Insert (Other): transcervical Foley catheter and an intravaginal dinoprostone controlled release insert
  Interventions: Drug: Cervidil 10 MG Vaginal Insert; Device: Foley Catheter
- Foley Catheter Alone (Other): a Foley catheter alone
  Interventions: Device: Foley Catheter

INTERVENTIONS:
Drug: Cervidil 10 MG Vaginal Insert — Dinoprostone vaginal insert is a thin, flat, polymeric slab which is rectangular in shape with rounded corners contained within the pouch of an off-white knitted polyester retrieval system, an integral part of which is a long tape. Each slab is buff colored, semitransparent and contains 10 mg of dinoprostone in a hydrogel insert. An integral part of the knitted polyester retrieval system is a long tape designed to aid retrieval at the end of the dosing interval or earlier if clinically indicated. The finished product is a controlled release formulation which has been found to release dinoprostone in vivo at a rate of approximately 0.3 mg/hr.
  Other Names: Dinoprostone
  Arms: Foley Catheter & Dinoprostone Insert
Device: Foley Catheter — The balloon on the end of the Foley catheter will be inflated with 30 mL of sterile water, pulled back against the internal os of the cervix, and taped to the maternal thigh under minimal tension.

SUMMARY:
In term women presenting for labor induction, combined use of the controlled release dinoprostone vaginal insert and Foley catheter for cervical ripening will decrease the median time from induction to vaginal delivery by at least four hours compared to the Foley catheter alone.

DETAILED DESCRIPTION:
Those who provide informed consent will be allocated by an online randomization system either to placement of a transcervical Foley catheter and an intravaginal dinoprostone controlled release insert or a Foley catheter alone. Randomization will be stratified by parity (nulliparous or parous).

In both study groups, the balloon on the end of the Foley catheter will be inflated with 30 mL of sterile water, pulled back against the internal os of the cervix, and taped to the maternal thigh under minimal tension. Also in both groups, the Foley catheter will be removed if any of the following occurs: 1) expulsion, 2) fetal heart rate tracing mandating evaluation for membrane rupture and placement of internal monitors, 3) spontaneous membrane rupture, or 4) if 12 hours has elapsed since placement. The dinoprostone insert will be removed if: 1) the fetal heart rate tracing mandates evaluation for membrane rupture and placement of internal monitors, 2) tachysystole develops (more than 5 contractions per 10 minutes averaged over 30 minutes, 3) spontaneous membrane rupture, or 4) 12 hours has elapsed since placement. Though these are the criteria for insert removal, in keeping with the pragmatic design of this trial, the decision regarding removal will be left to the discretion of the attending physician.

Women will remain recumbent for 30 minutes after agent placement and, except for trips to the restroom, will undergo continuous monitoring of uterine contractions and fetal heart rate. Oxytocin, according to standard intravenous protocol, will be allowed only after removal of cervical ripening agent(s). After specified cervical ripening, labor management will be at the discretion of the attending obstetrician, in keeping with the pragmatic nature of the study design.

Antibiotics will be administered if indicated for prophylaxis against early-onset neonatal infection with group B streptococci or for treatment of chorioamnionitis. Cesarean delivery will be performed, per the discretion of the attending obstetrician, for standard maternal or fetal indications.

Medical records will be reviewed no less than 30 days after delivery. Demographic, intrapartum, and outcome data will be entered into a computerized database.

ELIGIBILITY:
Inclusion Criteria:

1. Cervix ≤2 cm dilated; if 2 cm, <80% effaced
2. Gestational age 37 weeks or more
3. Singleton gestation
4. Cephalic presentation
5. Live fetus

Exclusion Criteria:

1. Contractions more frequent than every 5 minutes
2. Premature rupture of membranes
3. Prior uterine incision
4. Temperature 38C or higher
5. Fetal anomalies
6. Placenta previa
7. Suspected abruption or undiagnosed bleeding more than spotting
8. Fetal heart rate tracing prior to enrollment with no more than minimal variability, late decelerations, or more than two variable decelerations
9. HIV infection
10. Allergy to either latex or dinoprostone

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-09 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney K Edwards, MD, Principal Investigator — The University of Oklahoma Health Sciences Center
Locations (1):
- The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264

RESULTS

PARTICIPANT FLOW:
Groups:
- Nulliparous Foley Catheter & Dinoprostone Insert: patients with no prior pregnancies at or beyond 20 weeks who were randomized to have labor induction started with the dinoprostone insert and intracervical Foley catheter concurrently
- Nulliparous Foley Catheter Alone: patients with no prior pregnancies at or beyond 20 weeks who were randomized to have labor induction started with the intracervical Foley catheter alone
- Parous Foley Catheter & Dinoprostone Insert: patients with one or more prior pregnancies at or beyond 20 weeks who were randomized to have labor induction started with the dinoprostone insert and intracervical Foley catheter concurrently
- Parous Foley Catheter Alone: patients with one or more prior pregnancies at or beyond 20 weeks who were randomized to have labor induction with the intracervical Foley catheter alone
Period: Overall Study
Arm/Group | Nulliparous Foley Catheter & Dinoprostone Insert | Nulliparous Foley Catheter Alone | Parous Foley Catheter & Dinoprostone Insert | Parous Foley Catheter Alone
Started | 26 | 24 | 25 | 25
Completed | 26 | 24 | 25 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nulliparous Foley Catheter & Dinoprostone Insert | Nulliparous Foley Catheter Alone | Parous Foley Catheter & Dinoprostone Insert | Parous Foley Catheter Alone | Total
Number analyzed (Participants) | 26 | 24 | 25 | 25 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 25 | 25 | 100
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 25 | 25 | 100
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 13 | 11 | 8 | 44
  Black | 2 | 4 | 2 | 1 | 9
  Hispanic | 12 | 6 | 10 | 13 | 41
  Asian | 0 | 0 | 0 | 0 | 0
  Native American | 0 | 1 | 2 | 3 | 6
  Other | 0 | 0 | 0 | 0 | 0
Gestational age [Mean (Standard Deviation); unit: gestational age (weeks)] | 38.5 (1.5) | 38.9 (1.2) | 38.8 (1.3) | 38.9 (1.2) | 38.8 (1.3)
BMI [Mean (Standard Deviation); unit: body mass index] | 33 (1.5) | 35 (0.27) | 33.9 (6.8) | 34.8 (5.6) | 34.2 (3.4)
Chronic hyptertension [Count of Participants; unit: Participants] | 3 | 4 | 2 | 3 | 12
Diabetes [Count of Participants; unit: Participants] | 6 | 7 | 3 | 2 | 18
Preeclampsia [Count of Participants; unit: Participants] | 5 | 0 | 1 | 0 | 6
Gestational hypertension [Count of Participants; unit: Participants] | 5 | 9 | 8 | 1 | 23
Fetal growth restriction [Count of Participants; unit: Participants] | 1 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Median Times From Placement of Foley Catheter to Vaginal Delivery
Description: median time estimation for use of dinoprostone and foley catheter and foley catheter alone
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nulliparous Foley Catheter & Dinoprostone Insert | Nulliparous Foley Catheter Alone | Parous Foley Catheter & Dinoprostone Insert | Parous Foley Catheter Alone
Number analyzed (Participants) | 26 | 24 | 25 | 25
hours | 21.2 [16.6 to 38.0] | 31.3 [23.3 to 46.9] | 17.1 [13.6 to 21.9] | 14.8 [12.7 to 19.5]

2. Secondary Outcome: To Evaluate the Proportion of Patients That Delivered by 12 Hours and Proportion of Patients Delivered by 24 Hours
Description: To evaluate the proportion of patients that delivered vaginally by 12 hours and proportion of patients delivered vaginally by 24 hours.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Nulliparous Foley Catheter & Dinoprostone Insert | Nulliparous Foley Catheter Alone | Parous Foley Catheter & Dinoprostone Insert | Parous Foley Catheter Alone
Number analyzed (Participants) | 26 | 24 | 25 | 25
Participants
  Delivered vaginally by 12 hours | 2 | 1 | 3 | 6
  Delivered vaginally by 24 hours | 15 | 6 | 19 | 21

ADVERSE EVENTS:
Time Frame: adverse events data was collected beginning when the patient was randomized up until 30 days following delivery.
Arm/Group | Nulliparous Foley Catheter & Dinoprostone Insert | Nulliparous Foley Catheter Alone | Parous Foley Catheter & Dinoprostone Insert | Parous Foley Catheter Alone
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 4/24 | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 3/26 | 0/24 | 3/25 | 4/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nulliparous Foley Catheter & Dinoprostone Insert (N=26) | Nulliparous Foley Catheter Alone (N=24) | Parous Foley Catheter & Dinoprostone Insert (N=25) | Parous Foley Catheter Alone (N=25)
Superimposed preeclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Endometritis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nulliparous Foley Catheter & Dinoprostone Insert (N=26) | Nulliparous Foley Catheter Alone (N=24) | Parous Foley Catheter & Dinoprostone Insert (N=25) | Parous Foley Catheter Alone (N=25)
Neonatal ICU admission (Social circumstances) | 3 (3) | 0 (0) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Ferring shall have the right to review all clinical data arising from the research project. Sponsor/investigator shall provide any manuscript to Ferring prior to submission to permit at least 30 days for comment. Sponsor/investigator may incorporate the written suggestions or comments from Ferring in his/her own discretion. Ferring reserves the right to delay publication of clinical data arising from the research project, not to exceed 90 days to permit any intellectual property to be protected.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT03111316/Prot_SAP_000.pdf